CLINICAL TRIAL: NCT02992015
Title: A Clinical Trial Trial of Gemcitabine in Children with Newly-Diagnosed Diffuse Intrinsic Pontine Glioma (DIPG)
Brief Title: Gemcitabine in Newly-Diagnosed Diffuse Intrinsic Pontine Glioma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15-1621.cc
Record Dates: First submitted 2016-11-29; First posted 2016-12-14 (Estimated); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Diffuse Intrinsic Pontine Glioma
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine (Experimental): The entire therapy on this study is one dose of gemcitabine. No intrapatient dose modifications are necessary. Gemcitabine will be given at 2100 mg/m2 IV over 30 minutes within 4 hours of planned surgical procedure.
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine — Participants receive a one time IV dose of gemcitabine prior to having standard of care surgery.
  Other Names: Gemzar

SUMMARY:
Diffuse Intrinsic Pontine Glioma (DIPG) is an aggressive childhood brain tumor that, despite many past clinical trials, has never been shown to respond to chemotherapy. Radiation therapy (RT) is effective in extending life but is not curative; median overall survival is 11 months. It is still unclear why the hundreds of clinical trials involving chemotherapy of DIPG have failed to demonstrate any activity against the tumor. Given that many agents tried in clinical trials cross the blood brain barrier (BBB), it is possible that there are factors specific to DIPG and its location that prevent adequate drug penetration. Gemcitabine has been selected for this study because there is strong evidence of DIPG cell line inhibition in vitro and good BBB penetration. Furthermore, pediatric dosing and toxicity has been established in prior studies of children with relapsed solid tumors and leukemia.

The primary aim of this study is to determine the presence of gemcitabine in childhood DIPG tissue after systemic treatment with the drug. The secondary aim is to quantify the intratumoral gemcitabine concentration after systemic treatment.

Participants in this study will be given a one time IV dose of gemcitabine prior to having standard of care surgery. During surgery biopsies will be obtained for clinical and research purposes along with a blood sample. Because patients will be undergoing this biopsy as part of their standard of care therapy here at Children's Hospital Colorado, this is an optimal time to obtain a tumor biopsy for this study. The biopsy will serve to see if the study drug is penetrating the tumor. Patients will then enter a follow-up period for 30 days post surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 3 years and less than 18 years at the time of enrollment
2. Patients must meet both of the following:

   * Clinical findings consistent with a presumed new diagnosis of DIPG
   * Brain MRI findings consistent with a new diagnosis of DIPG in the opinion of the treating pediatric neuro-oncologist and neurosurgeon
3. Organ Function Requirements

   Adequate bone marrow function defined as:
   * Platelet count ≥100,000/µl (no platelet transfusion for more than 3 days)
   * Hemoglobin >8 g/dl and absolute neutrophil count (ANC) ≥1,000/µl

   Adequate coagulation defined as:
   * Prothrombin time (PT) and activated partial thromboplastin time (aPTT) ≤ upper limit of normal (ULN) for age.

   Adequate renal function defined as:
   * Creatinine clearane or radioisotope GFR > 70 ml/min/1.73 m2 or
   * Maximum serum creatinine (mg/dL) based on age/gender as follows:

     * Male 3 to <6 yrs: 0.8 mg/dL
     * Female 3 to <6 yrs: 0.8 mg/dL
     * Male 6 to <10 yrs: 1.0 mg/dL
     * Female 6 to <10 yrs: 1.0 mg/dL
     * Male 10 to <13 yrs : 1.2 mg/dL
     * Female 10 to <13 yrs: 1.2 mg/dL
     * Male 13 to <16 yrs: 1.5 mg/dL
     * Female 13 to <16 yrs: 1.4 mg/dL
     * Male 16 to <18 yrs : 1.7 mg/dL
     * Female 16 to <18 yrs: 1.4 mg/dL

   The threshold creatinine values in this Table were derived from the Schwartz formula for estimating GFR (Schwartz et al. J. Peds, 106:522, 1985) utilizing child length and stature data published by the CDC.

   Adequate liver function defined as:
   * Total bilirubin <3x ULN for age and SGOT (AST) and SGPT (ALT) <2.5x ULN for age
4. Patients must meet one of the following performance scores:

   * ECOG performance status scores of 0, 1, or 2;
   * Karnofsky score of ≥ 60 for patients > 16 years of age; or
   * Lansky score of ≥ 60 for patients ≤ 16 years of age
5. Pontine tumor biopsy is planned for the clinical care of the patient independent of study participation by the treating pediatric neurosurgeon and neuro-oncologist.
6. Informed consent and assent obtained as appropriate.

Exclusion Criteria:

1. Pregnant or breastfeeding patients due to teratogenic effects seen in animal/human studies.
2. Patients who have received any tumor-directed therapy prior to biopsy. Concurrent treatment with corticosteroids is allowed.
3. Patients with intratumoral hemorrhage larger than 0.5 cm on preoperative imaging.
4. Patients with personal or family history of bleeding disorders.
5. Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
PK testing levels of gemcitabine, its metabolite difluorodeoxyuridine (dFdU), and gemcitabine necleotides in peripheral blood and DIPG tissue | 2-12 hours post systemic admininstration of gemcitabine.
  The investigators will use liquid chromatography/tandem mass spectrometry (LC-MS/MS). An API 4000 instrument will be used, which has an approximate sensitivity of 0.1 ng/mg. Given the dimensions of the biopsy needle used, 10 mm length and 0.75 mm diameter, the investigators expect that each core will have an approximate volume of 4.5 mm2, which translates to a likely mass of 4.5 mg. Given that approximately 10 mg of tumor tissue has been necessary for quantification of gemcitabine and its matabolites in past studies, multiple cores of the six available for quantification from neighboring regions of the tumor may be combined; whenever possible. However, more than one separate measurement of concentrations will be done for each patient to determine any variation in concentrations across the tumor. An internal control measurement for gemcitabine will be determined using a variant gemcitabine compound enriched with 13C (Carbon 13).

CONTACTS AND LOCATIONS:
Overall Officials: Adam Green, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No